CLINICAL TRIAL: NCT02456181
Title: Investigation of the Efficacy of the JUMP Program of Mathematics Instruction
Brief Title: Investigation of Instructional Approaches to Elementary Math
Acronym: JUMP Math
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Rosemary Tannock, Senior Scientist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1000031586
Record Dates: First submitted 2015-05-25; First posted 2015-05-28 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Student Math Achievement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JumpMath (Experimental): The JUMP method focuses more on the mental activity involved in constructing mathematical knowledge. There is a strong emphasis on symbolic math (numbers, letters, mathematical symbols). Manipulatives are used prescriptively, in lessons carefully scaffolded to help students connect the objects (e.g., three buttons) to what they are intended to stand for (the magnitude "3").
  Interventions: Behavioral: JumpMath

INTERVENTIONS:
Behavioral: JumpMath

SUMMARY:
The overall aim of the proposed project is to test the efficacy of a relatively new, well-developed math program on the math achievement of elementary school students in mainstream classes in urban schools. Use of this program is increasing in Canada and the United Kingdom. Preliminary findings derived from uncontrolled trials and our own pilot, randomized controlled trial suggest it may yield meaningful gains in math achievement for both at-risk and achieving students, as indexed by their performance on national exams, in national math competitions, as well as on standardized measures of math achievement. However, the program has yet to be rigorously evaluated to determine its relative efficacy compared to the math programs typically used by school boards. The program provision of grade-specific teacher's guides and student workbooks (for grades 1 to 8), and minimal teacher training, points to its potential utility for full-scale implementation, should its efficacy be confirmed.

ELIGIBILITY:
Inclusion Criteria:

* The students must: have sufficient command of English to understand their teacher's instructions (as judged by their teacher, ELL students will be included provided they meet this criterion). They must have a signed parental consent form and also assent to participate in the study.

Exclusion Criteria:

* The students must have no uncorrected sensory, neurological, or physical impairments that would preclude the use of manipulatives, perceiving written math materials and figures, or hearing the teacher's instructions.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1156 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-08 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
The change scores on the Math Fluency, Calculation, and Applied Problems sub scales from a standardized battery (WJ-III) and on a curriculum based math measure, as well as on the results from a regional math assessment test. | Fall and Spring of School Years 1 and 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Solomon, PhD, Study Director — The Hospital for Sick Children
Locations (1):
- SickKids, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Solomon T, Dupuis A, O'Hara A, Hockenberry MN, Lam J, Goco G, Ferguson B, Tannock R. A cluster-randomized controlled trial of the effectiveness of the JUMP Math program of math instruction for improving elementary math achievement. PLoS One. 2019 Oct 30;14(10):e0223049. doi: 10.1371/journal.pone.0223049. eCollection 2019. PMID 31665143